CLINICAL TRIAL: NCT04748419
Title: Phase I/II Study Assessing Safety & Efficacy of Consolidative Hypofractionated Radiation Therapy for Boosting Residual Primary Lung Cancer With Durvalumab After Definitive Chemoradiation Therapy for Stage III Non-small Cell Lung Cancer
Brief Title: Safety & Efficacy of Consolidative Hypofractionated Radiation Therapy for Boosting Residual Lung Cancer With Durvalumab
Status: Active, not recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: University of Nebraska (Other)
Collaborators: AstraZeneca (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 0004-21-FB
Record Dates: First submitted 2021-02-05; First posted 2021-02-10 (Actual); Last update posted 2026-01-22 (Actual); Status verified 2025-11

CONDITIONS: Lung Cancer; Carcinoma, Non-Small Cell Lung
MeSH Terms: conditions — Lung Neoplasms; Carcinoma, Non-Small-Cell Lung | interventions — durvalumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (1):
- Hypofractionated radiation therapy (hfRT) with Durvalumab (Experimental): Combining consolidative radiation therapy (RT) using a hypofractionated regimen (hfRT) of 10Gy x 2 fractions for boosting the residual primary lung cancer with adjuvant anti-PD-L1 therapy (durvalumab), dose of 10 mg/kg infusion every two weeks concurrently for up to 12 months or disease progression.
  Interventions: Radiation: consolidative hypofractionated radiation therapy (hfRT); Drug: Durvalumab 50 MG/ML

INTERVENTIONS:
Radiation: consolidative hypofractionated radiation therapy (hfRT) — Consolidative hfRT will start from 6.5Gy x 2 fractions and dose escalate to 10Gy x 2 fractions in a 3+3 design
Drug: Durvalumab 50 MG/ML — Durvalumab 10 mg/kg via a 60-minute iv infusion every two weeks ± 3 days for up to 12 months
  Other Names: Imfinzi

SUMMARY:
This study is designed to determine if combining consolidative radiation therapy (RT) using a hypofractionated regimen (hfRT) (2 fractions) for boosting the residual primary lung cancer with adjuvant anti-PD-L1 therapy concurrently is safe and will provide better tumor control locoregionally and distantly than either modality alone.

DETAILED DESCRIPTION:
For safety reasons, consolidative hfRT will start from 6.5Gy x 2 fractions and dose escalate to 10Gy x 2 fractions in a 3+3 design. Consolidative hfRT will be delivered one to two months after finishing definitive chemoradiation therapy (dCRT) and concurrently with adjuvant anti-PD-L1 therapy using durvalumab in stage III non-small cell lung cancer (NSCLC).

At the final determined consolidative hfRT dose level, a total of thirty-two subjects with pathologically documented stage III NSCLC treated with dCRT will be enrolled for data analyses.

Follow-up assessments will occur every 3 months during durvalumab therapy for the first two years, then every 4-6 months after 2 years from study registration until confirmed disease progression or death. Primary endpoints include the safety of boost hfRT and concurrent anti-PD-L1 therapy adjuvantly following dCRT, and the 12-month progression-free survival to compare with historical results.

ELIGIBILITY:
Inclusion Criteria:

1. Pathologically diagnosed NSCLC (squamous cell carcinoma, adenocarcinoma, large- cell carcinoma, or non-small-cell lung cancer not otherwise specified), clinical stage III (AJCC 8th Ed.))
2. At time of consent, potential subjects must be a candidate for dCRT OR Must have received dCRT with at least 2 cycles of platinum-based chemotherapy concurrent with conventional fractionated radiation therapy with a total dose of 5700 - 6300 cGy
3. Patients must be aware of the nature of his/her disease and willingly provide written, informed consent. Including compliance with the requirements and restrictions listed in the informed consent form (ICF) and in this protocol. Written informed consent and any locally required authorization (e.g., Health Insurance Portability and Accountability Act in the US) obtained from the patient/legal representative prior to performing any protocol-related procedures, including screening evaluations.
4. Age > 19 years at time of study entry
5. Eastern Cooperative Oncology Group (ECOG) performance status of 0 or 1 at time of enrollment.
6. Life expectancy of > 12 weeks
7. Adequate normal organ and marrow function as defined below:

   * Hemoglobin ≥9.0 g/dL (5.59 mmol/L) (patients can be transfused to meet this criterion)
   * Absolute neutrophil count (ANC) > 1500 per mm3
   * Platelet count ≥100 x 109/L (>100,000 per mm3)
   * Serum bilirubin ≤1.5 x institutional upper limit of normal (ULN).
   * AST (SGOT)/ALT (SGPT) ≤2.5 x institutional upper limit of normal.
   * Calculated creatinine CL>40 mL/min by the Cockcroft-Gault formula
8. Evidence of post-menopausal status or negative serum pregnancy test for female pre-menopausal patients. Women will be considered post-menopausal if they have been amenorrheic for 12 months without an alternative medical cause.
9. Patient is willing and able to comply with the protocol for the duration of the study including undergoing treatment and scheduled visits and examinations including follow up

Exclusion Criteria:

1. Involvement in the planning and/or conduct of the study (applies to both AstraZeneca staff and/or staff at the study site)
2. Patients who have received prior anti-PD-1, anti PD-L1 or anti CTLA-4
3. Participation in another clinical study with an investigational product during the last 4 weeks
4. Concurrent enrolment in another clinical study, unless it is an observational (non- interventional) clinical study or during the follow-up period of an interventional study
5. Mixed small cell and non-small cell lung cancer histology
6. Patients who receive sequential chemoradiation therapy for locally advanced NSCLC
7. Patients with locally advanced NSCLC who have progressed during definitive platinum based, concurrent chemoradiation therapy
8. Any unresolved toxicity NCI CTCAE Grade >2 from previous anticancer therapy with the exception of alopecia, vitiligo, and the laboratory values defined in the inclusion criteria

   1. Patients with Grade ≥2 neuropathy will be evaluated on a case-by-case basis after consultation with the Study Physician.
   2. Patients with irreversible toxicity not reasonably expected to be exacerbated by treatment with durvalumab may be included only after consultation with the Study Physician. For example, post-operative neurological deficits for previous benign brain tumors, urinary incontinence from radical prostectomy for prostate cancer, peripheral neuropathy from chemotherapy for breast cancer.
9. Any concurrent chemotherapy, immunotherapy, biologic, or hormonal therapy for cancer treatment. Concurrent use of hormonal therapy for non-cancer-related conditions (e.g., hormone replacement therapy) is acceptable.
10. Major surgical procedure (as defined by the investigator) within 28 days to the first dose of immunotherapy (excluding the placement of vascular access) that would prevent administration of study drug or radiation therapy.
11. History of allogenic organ transplantation.
12. Active or prior documented autoimmune or inflammatory disorders within the past 2 years (including inflammatory bowel disease [e.g., colitis or Crohn's disease], diverticulitis [with the exception of diverticulosis], systemic lupus erythematosus, Sarcoidosis syndrome, or Wegener syndrome [granulomatosis with polyangiitis, Graves' disease, rheumatoid arthritis hypophysitis, uveitis, etc]). The following are exceptions to this criterion:

    1. Patients with vitiligo or alopecia
    2. Patients with hypothyroidism (e.g., following Hashimoto syndrome stable on hormone replacement or Graves' disease).
    3. Any chronic skin condition including psoriasis that does not require systemic therapy (within the past 2 years).
    4. Patients without active disease in the last 5 years may be included but only after consultation with the study physician.
    5. Patients with celiac disease controlled by diet alone.
13. Known allergy or hypersensitivity to Durvalumab or any excipient.
14. Uncontrolled intercurrent illness, including but not limited to, ongoing or active infection, symptomatic congestive heart failure, uncontrolled hypertension, unstable angina pectoris, cardiac arrhythmia, interstitial lung disease, serious chronic gastrointestinal conditions associated with diarrhea, or psychiatric illness/social situations that would limit compliance with study requirement, substantially increase risk of incurring AEs or compromise the ability of the patient to give written informed consent
15. History of another primary malignancy except for

    1. Malignancy treated with curative intent and with no known active disease ≥5 years before the informed consent and of low potential risk for recurrence
    2. Adequately treated non-melanoma skin cancer or lentigo maligna without evidence of disease
    3. Adequately treated carcinoma in situ without evidence of disease
16. History of primary immunodeficiency
17. Known history or active infection of tuberculosis, hepatitis B (known positive HBV surface antigen (HBsAg) result), hepatitis C, or human immunodeficiency virus (positive HIV 1/2 antibodies).
18. Current or prior use of immunosuppressive medication within 14 days before the first dose of durvalumab.

    1. Intranasal, inhaled, topical steroids, or local steroid injections (e.g., intra articular injection)
    2. Systemic corticosteroids at doses ≤10 mg/day of prednisone or its equivalent
    3. Steroids as premedication for hypersensitivity reactions (e.g., CT scan premedication)
    4. Systemic steroid administration required to manage toxicities arising from radiation therapy delivered as part of the chemoradiation therapy for locally advanced NSCLC is allowed.
19. Receipt of live attenuated vaccine within 30 days prior to the first dose of IP. Note: Patients, if enrolled, should not receive live vaccine whilst receiving IP and up to 30 days after the last dose of IP.
20. Female patients who are pregnant or breastfeeding or male or female patients of reproductive potential who are not willing to employ effective birth control from screening to 90 days after the last dose of durvalumab therapy.
21. Prior randomization or treatment in a previous durvalumab and/or tremelimumab clinical study regardless of treatment arm assignment.
22. Any prior Grade ≥3 immune-related adverse event (irAE) while receiving any previous immunotherapy agent, or any unresolved irAE >Grade 1.
23. Previous history of RT (other than RT as part of the dCRT for the current course of NSCLC) involving any part of lungs, chest wall, thoracic spine or breast(s).
24. Judgment by the investigator that the patient is unsuitable to participate in the study for any condition and the patient is unlikely to comply with study procedures, restrictions and requirements.
25. Mean QT interval corrected for heart rate using Fridericia's formula (QTcF) ≥470 ms calculated from 3 ECGs (2-5 minutes apart). Triplicate ECGs should only be performed if screening ECG shows QTcF ≥470 ms.

Min Age: 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 6 (Actual)
Dates: Start 2021-07-15 (Actual); Primary Completion 2026-03 (Estimated); Study Completion 2026-03 (Estimated)

PRIMARY OUTCOMES:
Evaluate the safety of combining hfRT and durvalumab by Adverse event assessed | 2 years
  Adverse events (AEs) will be assessed during the entire course of study
Evaluate progression free survival (PFS) when combining hfRT with adjuvant anti-PD-L1 therapy (durvalumab) | 12-month
  based on assessments according to RECIST 1.1

SECONDARY OUTCOMES:
Progression Free survival (PFS) when combining hfRT with adjuvant anti-PD-L1 therapy | 18 months
  PFS based on assessments according to RECIST 1.1a
Overall Survival hfRT and adjuvant anti-PD-L1 therapy | 12 months
  Overall Survival when combining hfRT with adjuvant anti-PD-L1 therapy

CONTACTS AND LOCATIONS:
Overall Officials: Chi Zhang, MD, PhD, Principal Investigator — University of Nebraska
Locations (1):
- University of Nebraska Medical Center, Omaha, Nebraska, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Coutu B, Lawrence E, Ganti AK, Marr A, Wichman C, Zhang C. Phase I/II study to evaluate consolidative hypofractionated radiation therapy for boosting the residual primary disease in combination with durvalumab after definitive chemoradiation therapy for stage III non-small cell lung cancer (NSCLC): study protocol for a prospective trial. J Thorac Dis. 2024 Jan 30;16(1):750-759. doi: 10.21037/jtd-23-304. Epub 2024 Jan 29. PMID 38410608

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2024-06-10): https://cdn.clinicaltrials.gov/large-docs/19/NCT04748419/Prot_SAP_000.pdf
  • Informed Consent Form (2025-11-03): https://cdn.clinicaltrials.gov/large-docs/19/NCT04748419/ICF_001.pdf